CLINICAL TRIAL: NCT04324424
Title: An Open-Label, Paralleled Study of the Pharmacokinetics of HMS5552 Following a Single Oral Dose in Renal Impaired Subjects and Matched Healthy Volunteers
Brief Title: A Clinical Study to Access the Pharmacokinetics of HMS5552 in Renal Impaired Subjects and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMM0110
Record Dates: First submitted 2020-03-23; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dorzagliatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Undialyzed ESRD subjects (P1) (Experimental): Part 1: Undialyzed end stage renal disease (ESRD) patients to receive a single dose of HMS5552 ( 25mg ) tablets orally
  .
  Interventions: Drug: HMS5552
- Healthy volunteers (H) (Experimental): Part 1: Matched healthy volunteers to receive a single dose of HMS5552 ( 25mg ) tablets orally
  Matching principle:
  H group and P1 group: 1:1 . The matched subjects should be in the same gender, age difference ±5 years, BMI difference ±15%
  Interventions: Drug: HMS5552
- Severe renal impaired subjects (P2) (Experimental): Part 2：Severe renal impaired subjects to receive a single dose of HMS5552 ( 25mg ) tablets orally
  Matching principle:
  P2 group and H group: 1:1 . The matched subjects should be in the same gender, age difference ±5 years, BMI difference ±15%
  Interventions: Drug: HMS5552
- Moderate renal impaired subjects (P3) (Experimental): Part 2：Moderate renal impaired subjects to receive a single dose of HMS5552 ( 25mg ) tablets orally
  Matching principle:
  P3 group and H group: 1:1 . The matched subjects should be in the same gender, age difference ±5 years, BMI difference ±15%
  Interventions: Drug: HMS5552
- Mild renal impaired subjects (P4) (Experimental): Part 2：Mild renal impaired subjects to receive a single dose of HMS5552 ( 25mg ) tablets orally
  Matching principle:
  P4 group and H group: 1:1 . The matched subjects should be in the same gender, age difference ±5 years, BMI difference ±15%
  Interventions: Drug: HMS5552

INTERVENTIONS:
Drug: HMS5552 — single dose of HMS5552 25mg

SUMMARY:
The objectives of this study is to access the pharmacokinetics and safety of HMS5552 in single dose in renal impaired subjects and matched healthy adult subjects.

DETAILED DESCRIPTION:
This is an open-label and paralleled study with single oral dose of HMS5552 given to renal impaired subjects and body index matched healthy volunteers.

The primary objective is to access the pharmacokinetic profiles of HMS5552 in 25 mg dose in renal impaired subjects and (gender, age and BMI) matched healthy adult subjects.

The secondary objective is to characterize the safety profiles of HMS5552 in single dose in renal impaired subjects.

The subjects include ESRD subjects without dialysis (P1 group), severe (P2 group), moderate (P3 group), mild (P4 group), and healthy subjects (H Group) matched with renal impairment subjects in gender, age and BMI. The number of subjects in each group was 6-8.

The study is divided into two parts:

* Part 1: ESRD subjects without dialysis and matched healthy subjects (P1 and H groups; n = 8 for each group);
* Part 2: subjects with severe, moderate and mild renal impairment (P2, P3 and P4 groups; n = 6-8 in each group).

The study initiates from Part 1. The data will be evaluated at the end of Part 1 as the medium term. Compared with the matched healthy subjects, if the mean AUC of HMS5552 (either AUClast or AUCinf) increased by ≥ 100% in ESRD subjects without dialysis, which means Part 2 will need to be conducted. The process of Part 2 is the same as that of Part 1

ELIGIBILITY:
Inclusion Criteria:

* For renal impaired subjects:

  1. Male and female subjects between ages of 18 and 65 years, no less than 3 subjects in each gender.
  2. Body weight≥50kg for male and ≥45kg for female； BMI: 18.5~30 kg/m2
  3. eGFR: P1 < 15 mL/min/1.73 m2；P2: 15～29 mL/min/1.73 m2；P3: eGFR 30～59 mL/min/1.73 m2；P4: 60～89 mL/min/1.73 m2，and ACR≥ 3 mg/mmol；
  4. Normal physical conditions, vital signs,12 lead ECG and laboratory recording, blood potassium 3.5~5.5mmol/L;
  5. Left ventricular ejection fraction (LVEF) ≥50%
  6. Willing to sign the informed consent form (ICF) and take reliable contraceptive measures within 6 months after taking the last dose of study drug;
  7. Willing to adhere to the protocol requirement.
* For healthy volunteers:

  1. Male and female subjects between ages of 18 and 65 years, no less than 3 subjects in each gender.
  2. Body weight≥50kg for male and ≥45kg for female； BMI: 18.5~30 kg/m2
  3. MDRD eGFR: ≥90 mL/min/1.73 m2；
  4. Gender, age (±5 years) and BMI (±15%) matched with corresponding subject in P1 group
  5. Normal physical conditions, vital signs,12 lead ECG and laboratory recording
  6. Systolic pressure: 90～140 mmHg，diastolic pressure:50～90 mmHg；
  7. Willing to sign the informed consent form (ICF) and take reliable contraceptive measures within 6 months after taking the last dose of study drug;
  8. Willing to adhere to the protocol requirement.

Exclusion Criteria:

* Subjects with impaired renal function cannot be enrolled if they meet one of the following criteria:

  1. Acute renal failure;
  2. History of allergy;
  3. In addition to renal impaired function, investigators adjudicate subjects have diseases that may affect drug absorption, distribution, metabolism or excretion;
  4. Any other disease may receive treatment or surgery during the study
  5. Abnormal of ECG performance or laboratory recording;
  6. Family history of QT prolongation syndrome;
  7. Have unstable cardiovascular disease, lung disease, gastrointestinal disease, liver disease, blood disease, mental disease, nervous system disease, immune deficiency disease or any malignant tumor;
  8. History of cardiovascular and cerebrovascular disease;
  9. Hear failure (NYHA) class III or IV;
  10. Severe anemia, CHC<6.0g/dl at screening;
  11. Severe infection, trauma, gastrointestinal operation or other surgery within 4 weeks before screening;
  12. History of a) Type 1 diabetes, b) Acute complications of diabetes;
  13. Serious hypoglycemia events within 3 months before screening;
  14. More than 5 cigarettes per day within 3 months before screening;
  15. Alcohol addicts;
  16. History of drug abuse;
* Healthy subjects cannot be enrolled if they meet one of the following criteria:

  1. History of allergy;
  2. Investigators adjudicate subjects have diseases that may affect drug absorption, distribution, metabolism or excretion;
  3. Any other disease may receive treatment or surgery during the study
  4. Abnormal of ECG performance or laboratory recording;
  5. Family history of QT prolongation syndrome;
  6. Have unstable cardiovascular disease, lung disease, gastrointestinal disease, liver disease, blood disease, mental disease, nervous system disease, immune deficiency disease or any malignant tumor; history of cardiovascular and cerebrovascular disease within 6 months before screening; severe infection, trauma, gastrointestinal operation or other surgery within 4 weeks before screening;
  7. Anemia caused by any reason;
  8. History of hypoglycemia (<3.9mmol/L);
  9. More than 5 cigarettes per day within 3 months before screening;
  10. Alcohol addicts;
  11. History of drug abuse;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of Cmax | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of AUClast | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of AUCinf | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.

SECONDARY OUTCOMES:
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of Cmax,u (if applicable) | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of AUClast,u (if applicable) | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of AUCinf,u (if applicable) | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of Tmax (if applicable) | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of T1/2 (if applicable) | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of CL/F (if applicable) | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of Vz/F (if applicable) | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of fu (if applicable) | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of Ae (if applicable) | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of CLr (if applicable) | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Miao, MD, Principal Investigator — West China Hospital; Ping Fu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miao J, Fu P, Ren S, Hu C, Wang Y, Jiao C, Li P, Zhao Y, Tang C, Qian Y, Yang R, Dong Y, Rong J, Wang Y, Jin X, Sun Y, Chen L. Effect of renal impairment on the pharmacokinetics and safety of dorzagliatin, a novel dual-acting glucokinase activator. Clin Transl Sci. 2022 Feb;15(2):548-557. doi: 10.1111/cts.13174. Epub 2021 Nov 11. PMID 34706161